CLINICAL TRIAL: NCT03922191
Title: Post-Surgical Mediastinitis: Retrospective Study of Cases Treated Within the CHU Brugmann Hospital
Brief Title: Post-Surgical Mediastinitis Within the CHU Brugmann Hospital
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Medical Director of the Hospital, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Pauels
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Mediastinitis
MeSH Terms: conditions — Mediastinitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric population: Infants diagnosed with cardiac post-surgery mediastinitis within the HUDERF Hospital within the last 20 years.
  Interventions: Other: Data extraction from medical files
- Adult population: Adults diagnosed with cardiac post-surgery mediastinitis within the CHU Brugmann Hospital within the last 20 years.
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Mediastinitis is an infectious complication that can occur after cardiac surgery. The incidence varies between 1 and 3% depending on the type of procedure and the patient's condition. The mortality of this severe postoperative complication rises from 10 to 35%, which makes it dreadful.

The major risk factors reported are obesity, diabetes, and immunosuppressive therapy. There are other less important ones: age, coronary bypass grafting (especially if using the two internal mammary arteries), nosocomial pneumonia, dialysis, prolonged mechanical ventilation, long operative asepsis, undrained retro-sternally hematoma, prolonged pre-operative hospitalization...).

Prevention is very important. The principle of asepsis must absolutely be respected. The use of prophylactic antibiotic therapy is recommended.

The most commonly encountered organisms are Staphylococcus aureus, coagulase-negative Staphylococci and gram-negative bacilli.

There are several treatment modalities that vary between centers and may be different depending on the surgical team's experience and the depth or extent of the infection. The common principles of these treatments are: antibiotic therapy and surgical debridement (the timing of which may vary). The timing and modalities of wound closure are subject to variations: immediate sternal closure with placement of multiple or delayed drains. Muscle flaps or large omentum transplant may be necessary if tissue loss is too important.

The investigators propose to review their experience in the treatment of cardiac post-surgery mediastinitis at Brugmann University Hospital in the last 20 years in both adult and pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* post-cardiac surgery mediastinitis
* patients of the CHU Brugmann (adults) and HUDERF (pediatric) Hospitals

Exclusion Criteria:

- none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the CHU Brugmann (adults) and HUDERF (pediatric) Hospitals, treated for post-cardiac surgery mediastinitis.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Duration of the hospitalization | 20 years
  Duration of the hospitalization
Mortality at six months | 6 months
  Mortality rate six months after mediastinitis diagnosis
Percentage of recurrence | 20 years
  Percentage of recurrence of mediastinitis
Percentage of re-hospitalization | 20 years
  Percentage of re-hospitalizations caused by mediastinitis
Duration of the antibiotic treatment | 20 years
  Duration of the antibiotic treatment for mediastinitis
Presence of superinfection | 20 years
  Presence of superinfection

SECONDARY OUTCOMES:
Date of birth | 20 years
  Demographic data : Date of birth.
Sex | 20 years
  Demographic data : sex.
Risk factors | 20 years
  Demographic data : presence of risk factors (obesity, diabetes...).
Surgical intervention | 20 years
  Name of the surgical intervention that caused the mediastinitis
Germ identification | 20 years
  Name of the germ causing the mediastinitis
Type of treatment | 20 years
  Name of the antibiotics used to treat the mediastinitis

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pauels, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No